CLINICAL TRIAL: NCT05055661
Title: Pragmatic Study of the Effectiveness of Pharmaceutical Teleconsultation in Adults With Asthma
Brief Title: Pharmaceutical Teleconsultation in Adults With Asthma
Acronym: EPETEFAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Stella Pegoraro Alves Zarpelon, PhD candidate, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UFRGS EPETEFAS
Record Dates: First submitted 2021-09-03; First posted 2021-09-24 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Asthma
Keywords: Pragmatic Clinical Trial; Pharmaceutical Services; Telemedicine
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (No Intervention): Patients randomized to the control group will receive health education, audiovisual educational meterial regarding the use of inhalers and inhalators spacers and be contacted throughout the six months to collect the study variables, by telephone contact.
- The intervention group (Experimental): Patients randomized to the intervention grop will receive the same health education as the control group at the reference Basic Health Unit and also will be carried, once a month, the pharmaceutical teleconsultation during six months, by video call. The study variables will be collected in the same periods as the control group patients, by telephone contact.
  Interventions: Other: Pharmaceutical Teleconsultation

INTERVENTIONS:
Other: Pharmaceutical Teleconsultation — The pharmacist will apply the teleconsultation according to the elaborated workflows and will follow in seven steps: scheduling the teleconsultation; pre-consultation, in which the pharmacist will make a checklist of the adequacy of the teleconsultation environment; presentation of the professional and the objectives of the teleconsultation to the patient; search for information about the patient and their pharmacotherapy; identification of problems related to pharmacotherapy; elaboration of a care plan and appointment for the re-consultation.
  Arms: The intervention group

SUMMARY:
The investigators propose a pragmatic randomized clinical study, consisting of two groups, the control group with health education and the intervention group with teleconsultation. The research team comprises pharmacists, students, and professors who work in a pharmaceutical service of secondary health care linked to the public university. The investigators will conduct the study exclusively remotely, following the patients for six months. The research team will implement and structure an ambiance to adapt the face-to-face pharmaceutical consultation into the pharmaceutical teleconsultation. The evaluated outcomes, in both groups, will be the scores of the Asthma Control Test, the Asthma Quality of Life, and the hospitalization rate and admission to urgency/emergency services.

DETAILED DESCRIPTION:
It is a pragmatic, randomized, single-blind clinical trial based on a population of users diagnosed with asthma, registered in the Pharmaceutical Assistance Network in Porto Alegre (Rio Grande do Sul, Brazil). The study will be conducting exclusively by remote means, in the premises of the Collaborating Center for Pharmaceutical Services (CECOL-FAR), belonging to the Faculty of Pharmacy of the Federal University of Rio Grande do Sul (UFRGS). Characterized as a pharmaceutical service of secondary care, the CECOL-FAR/UFRGS, in the pre-pandemic COVID-19, used to provide assistance in face-to-face pharmaceutical consultations to patients who did not adhere to the asthma treatment.

The research team of the study, composed of pharmacists from CECOL-FAR/UFRGS, students and professors of the Postgraduate degree in Pharmaceutical Services (PPGASFAR) at UFRGS, will restructure and adapt the face-to-face pharmaceutical consultation for teleconsultation, with the creation of work processes, elaboration of research flows and standard operating procedures (SOP).

The pilot study, carried out through simulated situations, will evaluate these new practices regarding the processes' suitability, feasibility, and scope. After the pilot project adaptation, the documents will be applied to the study in the implementation of pharmaceutical teleconsultation.

Study participants will be drawn from the population of users diagnosed with asthma treated in Primary Health Care. The physician will apply the Asthma Control Test (ACT) to assess the control of asthma symptoms. For patients considered to have uncontrolled asthma, it will be verified whether it meets the other eligibility criteria for inclusion in the study. If the criteria are met, individuals will be referred for care at CECOL-FAR, via the system of regulation of specialized consultations of the Unified Health System (SUS), after medical consultation.

Once scheduled in the system, the research team will contact the patient via telephone and offer two types of service: pharmaceutical consultation, in which the patient must travel to CECOL-FAR on a date and time scheduled for face-to-face consultation or teleservice. Patients who opt for telecare will be invited to participate in the study.

Patients considered for the study must meet the following inclusion criteria: diagnosis of asthma, age equal to or greater than 18 years old, ACT scores below 20 points, agree to participate in the teleservice and acceptance by written or audio message, from the informed consent. Patients who do not attend the research team in the foreseen contacts and patients with cognitive problems will be excluded from the study.

Patients will be randomized, using specific software, to one of two groups: control group (Health education) or intervention group (Pharmaceutical teleconsultation). The research team will accompany the participants of both groups for six months by remote, telephone contact, and video call, using Google Meet® or Whatsapp®.

The population considers all patients diagnosed with asthma followed at the municipal primary health care network. Thus, the patient sample size needed to obtain 1-α = 0.95 confidence, and ε = 7% maximum error was estimated for a minimum of 196 patients (98 patients in each group), estimating 80% power to detect a difference of 0.1 between the proportion of the null hypothesis and the alternative hypothesis. With expected losses of 25%, the sample was increased to 123 individuals in each group, totaling 246 patients.

The chi-square test for categorical variables and the t-student test for continuous characteristics will be applied to compare the baseline characteristics between control and intervention groups. The variables compared will be related to the clinical and humanistic outcomes observed, based on the ACT score, indicating the effective control of asthma. The hypothesis tests will identify significant differences between individuals for the analysis of results, adopting a significance level of 0.05. Data analysis will follow an intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma;
* Age equal to or greater than 18 years;
* ACT score less than 20 points;
* Patients who can read and write;
* Possibility of using the WhatsApp® application (by video call)
* Acceptance by written or audio message, from the informed consent.

Exclusion Criteria:

* Patients who do not attend the research team in the foreseen contacts, always in five attempts for each stage of the study, whether via telephone contact or video calls, will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change from Asthma Control test (ACT) score at 6 months | Applied in three moments: in beginning of the study, month 3, and month 6
  The ACT is an important marker of the severity of the disease and parameter for determining the need to adjust the treatment plan.
Hospitalization rate and admissions to urgency/emergency services | Collected at the end of the study (month 6)
  The data will be made available by the Municipal Health Department

SECONDARY OUTCOMES:
Change from Asthma Quality of Life Questionnaire (AQLQ) values at 6 months | Applied in two moments: in the beginning of the study and month 6
  Self-applicable, sent to patients by online form.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Bueno, PhD, Principal Investigator — Federal University of Rio Grande do Sul; Stella Pegoraro Alves Zarpelon, MSc, Study Director — Federal University of Rio Grande do Sul; Diogo Pilger, PhD, Study Director — Federal University of Rio Grande do Sul; Aline de Lima Nogare, MSc, Study Chair — Federal University of Rio Grande do Sul; Luiza Fedatto Vidal, BSc, Study Chair — Federal University of Rio Grande do Sul; Fernando Kreutz, PhD, Study Chair — Federal University of Rio Grande do Sul; Luciane Piva Klein, BSc, Study Chair — Federal University of Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pizzichini MMM, Carvalho-Pinto RM, Cancado JED, Rubin AS, Cerci Neto A, Cardoso AP, Cruz AA, Fernandes ALG, Blanco DC, Vianna EO, Cordeiro Junior G, Rizzo JA, Fritscher LG, Caetano LSB, Pereira LFF, Rabahi MF, Oliveira MA, Lima MA, Almeida MB, Stelmach R, Pitrez PM, Cukier A. 2020 Brazilian Thoracic Association recommendations for the management of asthma. J Bras Pneumol. 2020 Mar 2;46(1):e20190307. doi: 10.1590/1806-3713/e20190307. eCollection 2020. PMID 32130345
- [Background] Erdmann AL, de Andrade SR, de Mello AL, Drago LC. Secondary health care: best practices in the health services network. Rev Lat Am Enfermagem. 2013 Jan-Feb;21 Spec No:131-9. doi: 10.1590/s0104-11692013000700017. English, Portuguese. PMID 23459900
- [Background] Alexander E, Butler CD, Darr A, Jenkins MT, Long RD, Shipman CJ, Stratton TP. ASHP Statement on Telepharmacy. Am J Health Syst Pharm. 2017 May 1;74(9):e236-e241. doi: 10.2146/ajhp170039. No abstract available. PMID 28438829
- [Background] Niznik JD, He H, Kane-Gill SL. Impact of clinical pharmacist services delivered via telemedicine in the outpatient or ambulatory care setting: A systematic review. Res Social Adm Pharm. 2018 Aug;14(8):707-717. doi: 10.1016/j.sapharm.2017.10.011. Epub 2017 Oct 28. PMID 29100941
- [Background] Parreiras Martins MA, Fonseca de Medeiros A, Dias Carneiro de Almeida C, Moreira Reis AM. Preparedness of pharmacists to respond to the emergency of the COVID-19 pandemic in Brazil: a comprehensive overview. Drugs Ther Perspect. 2020;36(10):455-462. doi: 10.1007/s40267-020-00761-7. Epub 2020 Jul 31. PMID 32837194
- [Background] Coutinho Eda S, Huf G, Bloch KV. [Pragmatic clinical trials: an option in the construction of health-related evidence]. Cad Saude Publica. 2003 Jul-Aug;19(4):1189-93. doi: 10.1590/s0102-311x2003000400039. Epub 2003 Sep 8. Portuguese. PMID 12973582
- [Background] Juniper EF, Guyatt GH, Epstein RS, Ferrie PJ, Jaeschke R, Hiller TK. Evaluation of impairment of health related quality of life in asthma: development of a questionnaire for use in clinical trials. Thorax. 1992 Feb;47(2):76-83. doi: 10.1136/thx.47.2.76. PMID 1549827
- [Background] Franco R, Nascimento HF, Cruz AA, Santos AC, Souza-Machado C, Ponte EV, Souza-Machado A, Rodrigues LC, Barreto ML. The economic impact of severe asthma to low-income families. Allergy. 2009 Mar;64(3):478-83. doi: 10.1111/j.1398-9995.2009.01981.x. Epub 2009 Feb 6. PMID 19210355
- [Background] Nathan RA, Sorkness CA, Kosinski M, Schatz M, Li JT, Marcus P, Murray JJ, Pendergraft TB. Development of the asthma control test: a survey for assessing asthma control. J Allergy Clin Immunol. 2004 Jan;113(1):59-65. doi: 10.1016/j.jaci.2003.09.008. PMID 14713908
- [Background] Roxo JP, Ponte EV, Ramos DC, Pimentel L, D'Oliveira Junior A, Cruz AA. [Portuguese-language version of the Asthma Control Test]. J Bras Pneumol. 2010 Mar-Apr;36(2):159-66. doi: 10.1590/s1806-37132010000200002. Portuguese. PMID 20485935
- See also: Global Initiative for Asthma. Global Strategy for Asthma Management and Prevention — http://ginasthma.org/wp-content/uploads/2021/05/GINA-Main-Report-2021-V2-WMS.pdf
- See also: Brazil, Ministry of Health. Resolution No. 466. Provides for guidelines and regulatory standards for research involving human beings — https://bvsms.saude.gov.br/bvs/saudelegis/cns/2013/res0466_12_12_2012.html.
- See also: General Law for the Protection of Personal Data (LGPD), Brazil — http://www.planalto.gov.br/ccivil_03/_ato2015-2018/2018/lei/l13709.htm
- See also: Brazil, Ministry of Health. Circular Letter No. 2. Guidelines for research procedures at any stage in a virtual environment — http://conselho.saude.gov.br/images/Oficio_Circular_2_24fev2021.pdf